CLINICAL TRIAL: NCT05081076
Title: Health of Peri-implant Tissues Adjacent to Glazed or Polished Zirconia Surface: a Randomized, Intra-subject, Clinical Trial
Brief Title: Health of Peri-implant Tissues Adjacent to Zirconia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidade Católica do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: CAAE 45255621.2.0000.5336
Record Dates: First submitted 2021-09-14; First posted 2021-10-18 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Peri-Implantitis
Keywords: monolithic zirconia; dental implants; peri-implant tissues; surface finishing
MeSH Terms: conditions — Peri-Implantitis | interventions — Dental Polishing

STUDY DESIGN:
Intervention Model Description: The study design is a randomized, prospective, paired, clinical trial with intra-subject comparison. Each zirconia crown to be placed over the dental implant has two sides (mesial and distal), which will receive a randomised surface finishing treatment in the laboratory fabrication procedure.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomisation of surface finishing treatment per side (mesial or distal) of each zirconia crown will be made at the laboratory fabrication step, and the treatment codes will be known only by the certified technician and Projec PI. The clinician, who is also the investigator and outcomes assessor, will not assess the codes until the final data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glazed surface (Active Comparator): One side of the zirconia crown will receive glazed surface treatment according to standard laboratory procedure and manufacturer's recommendations (Ceramill Stain & Glaze Kit).
  Interventions: Device: Glazing
- Polished surface (Experimental): The contralateral side of the zirconia crown will receive polished surface treatment (polishing rubbers kit in the sequence indicated by the manufacturer - EVE DIACERA Finishing and Polishing Kit, EVE Ernst Vetter GmbH - Germany).
  Interventions: Device: Polishing

INTERVENTIONS:
Device: Glazing — The zirconia surface will be submitted to a vitrification procedure (glazing) in a specific ceramic oven using the Ceramill Stain & Glaze Kit, following the manufacturer's instructions.
  Arms: Glazed surface
Device: Polishing — The zirconia surface will be submitted to a polishing procedure using a polishing rubbers kit in the sequence indicated by the manufacturer (EVE DIACERA Finishing and Polishing Kit, EVE Ernst Vetter GmbH - Germany).
  Arms: Polished surface

SUMMARY:
Background: The control and maintenance of implants, bone tissue and soft tissue are fundamental for the clinical success of implant prostheses (PSIs). The type of ceramic surface finish can modify the biological response of peri-implant tissues adjacent to PSIs over time.

Objective: To prospectively assess whether the peri-implant health of soft and hard tissues adjacent to monolithic zirconia PSIs varies with the type of surface finish (glazed or polished). It will also be evaluated if the patient perceives any clinical, comfort or satisfaction difference.

Methodology: The study design is a randomized, prospective, paired clinical trial, with intra-subject comparison. The sample will consist of consecutive patients in need and indication for treatment with monolithic zirconia PSIs, attended at the Military Policlinic of Porto Alegre and in a private practice by a single specialist researcher. For each PSI, the allocation of a glazed or polished surface in contact with the soft gingival tissue will be randomized on the mesial and distal sides of the crown. Data will be collected by routine clinical and radiographic examination with a focus on peri-implant health (hygiene index, gingival bleeding index, crestal bone level), satisfaction questionnaire and intraoral images (thermography and photographs), after one week of installation of the PSI and in six months, one year and two years. The data will be analyzed by descriptive and inferential statistics, at the significance level of 0.05.

DETAILED DESCRIPTION:
The control and maintenance of implant, bone and soft tissue are fundamental for the clinical success of prostheses over implants (PSIs). The type of ceramic surface finish can modify the biological response of peri-implant tissues adjacent to PSIs over time.

AIM To prospectively assess whether the peri-implant health of soft and hard tissue adjacent to monolithic PSIs varies with the type of surface finish (glazed or polished).

METHODS The study design is a randomized, prospective, paired, clinical trial with intra-subject comparison, and the research protocol will follow the Resolution 466/12 of the Brazilian National Health Council and the Declaration of Helsinki.

Sample A non-probabilistic sample will consist of consecutive patients in need of treatment with unitary PSIs made of monolithic zirconia, being attended at the Military Polyclinic of Porto Alegre and in a private practice by the same specialist researcher (DBS). Patients will be selected according to the eligibility criteria.

Sample size calculation: In the systematic review of Linkevicius and Vaitelis (2015) on the effect of zirconia or titanium abutments on peri-implant tissues, the 11 clinical studies included for biological outcomes had samples from 11 to 81 patients, with 11 to 45 abutments. In a total of 145 zirconia abutments, 12 (8.2%) had biological complications. There is no current clinical studies on glaze and PSI polishing in monolithic zirconia and outcomes of peri-implant health. So, a priori, the initial sample will consist of 30 PSIs (30 pairs to be compared: Glaze vs. Polishing). The definitive sample size will be calculated after preliminary data analysis from the initial six months of data collection.

PSIs crowns will be made on metallic abutments (Variobase or Anatomic Abutment, Straumann) and milled in monolithic zirconia (Amann Girrbach, Austria), using a CAD/CAM technique with molding or intra-oral scanning and in-lab milling. For each PSI, the mesial and distal faces will receive one experimental treatment (surface finishing) at random, to be defined by drawing lots: glazed surface treatment (Ceramill Stain & Glaze Kit), or polished surface treatment (polishing rubbers kit in the sequence indicated by the manufacturer - EVE DIACERA Finishing and Polishing Kit, EVE Ernst Vetter GmbH - Germany).

All PSIs will be installed according to standardized clinical protocol in the routine of dental clinics where the patients will be seen. After installing the PSI, the clinical data will be collected by clinical-radiographic exam and photographs at the following times: after one week of installation of the PSI (T0 - baseline) and in six months (T1), one year (T2) and two years (T3) of follow-up.

Clinical-radiographic Examination A single trained examiner (D.B.S.) will carry out the collection of clinical and radiographic data for each PSI installed through non-invasive procedures already used in dentistry.

In the clinical exam the following aspects will be evaluated on each face (glazed or polished) of the PSI:

* Hygiene Index: will be visually evaluated the presence of bacterial plaque (biofilm) and the presence of visible inflammation.
* Index of Gingival Bleeding: Gingival probe around the zirconia crown, as per the last consensus of Periodontics (Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions).
* Patient Satisfaction: a 100-mm visual analogue scale will be used
* Infrared thermography
* Radiographic evaluation for peri-implant levels analysis (potential bone loss)

Statistical analysis The data will be analyzed by descriptive and inferential statistics (alpha = 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Healing time of at least two months for patients who underwent extraction in areas to be rehabilitated with implants
* Adequate bone volume at the implant site (ie, sufficient for placement of an implant of at least 3.3 mm in diameter and 6 mm in length) assessed by preoperative CT and clinical evaluation.
* Use of Straumann bone level or conical bone level implants, with NC or RC platforms.

Exclusion Criteria:

* Patients with systemic diseases (e.g., heart disease, leukocyte and coagulation disorders, metabolic disorders, immunosuppression)
* History of radiotherapy in the head and neck region
* Current treatment with steroids and/or bisphosphonates
* Neurological or psychiatric impairment that can interfere with good oral hygiene
* Smoking (more than 10 cigarettes a day)
* History of illicit drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline Hygiene Index at six months | from one week of installation of the PSI (T0 - baseline) to six months (T1) of follow-up
  Hygiene Index: will be visually evaluated the presence of bacterial plaque (biofilm) and the presence of visible inflammation
Change from six-month Hygiene Index at one year | from six months (T1) to one year (T2) of follow-up
  Hygiene Index: will be visually evaluated the presence of bacterial plaque (biofilm) and the presence of visible inflammation
Change from one-year Hygiene Index at two years | from one year (T2) to two years (T3) of follow-up
  Hygiene Index: will be visually evaluated the presence of bacterial plaque (biofilm) and the presence of visible inflammation
Change from baseline Index of Gingival Bleeding at six months | from one week of installation of the PSI (T0 - baseline) to in six months (T1) of follow-up
  Index of Gingival Bleeding: Gingival probe around the zirconia crown, as per the last consensus of Periodontics (Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions)
Change from six-month Index of Gingival Bleeding at one year | from six months (T1) and one year (T2) of follow-up
  Index of Gingival Bleeding: Gingival probe around the zirconia crown, as per the last consensus of Periodontics (Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions)
Change from one-year Index of Gingival Bleeding at two years | from one year (T2) to two years (T3) of follow-up
  Index of Gingival Bleeding: Gingival probe around the zirconia crown, as per the last consensus of Periodontics (Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions)

SECONDARY OUTCOMES:
Change in baseline Overal Satisfaction at six months | from one week of installation of the PSI (T0 - baseline) to in six months (T1) of follow-up
  Patient Satisfaction: a 100-mm visual analogue scale will be used
Change in six-month Overal satisfaction at one year | from six months (T1) to one year (T2) of follow-up
  Patient Satisfaction: a 100-mm visual analogue scale will be used
Change in one-year Overal satisfaction at two years | from one year (T2) to two years (T3) of follow-up
  Patient Satisfaction: a 100-mm visual analogue scale will be used
Change in baseline Infrared thermography score at six months | from one week of installation of the PSI (T0 - baseline) to six months (T1) of follow-up
  Infrared termograms obtained from a portable infrared camera will be assessed with the dedicated software to obtain a score measure of each region of interest after calibration procedures
Change in six-month Infrared thermography score at one year | from six months (T1) to one year (T2) of follow-up
  Infrared termograms obtained from a portable infrared camera will be assessed with the dedicated software to obtain a score measure of each region of interest after calibration procedures
Change in one-year Infrared thermography score at two years | from one year (T2) to two years (T3) of follow-up
  Infrared termograms obtained from a portable infrared camera will be assessed with the dedicated software to obtain a score measure of each region of interest after calibration procedures
Change in baseline Bone loss at six months | from one week of installation of the PSI (T0 - baseline) to six months (T1) of follow-up
  Radiographic images will be analysed with a specific software for peri-implant level measurements at the vertical implant axis, at the mesial and distal sides
Change in six-month Bone loss at one year | from six months (T1) to one year (T2) of follow-up
  Radiographic images will be analysed with a specific software for peri-implant level measurements at the vertical implant axis, at the mesial and distal sides
Change in one-year Bone loss at two years | from one year (T2) to two years (T3) of follow-up
  Radiographic images will be analysed with a specific software for peri-implant level measurements at the vertical implant axis, at the mesial and distal sides

CONTACTS AND LOCATIONS:
Overall Officials: Rosemary SA Shinkai, DDS, PhD, Study Chair — Pontificia Universidade Católica do Rio Grande do Sul (PUCRS)
Locations (1):
- Pontificia Universidade Católica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No
IPD may be shared with other researchers upon justified request.

REFERENCES:
- [Background] Linkevicius T, Vaitelis J. The effect of zirconia or titanium as abutment material on soft peri-implant tissues: a systematic review and meta-analysis. Clin Oral Implants Res. 2015 Sep;26 Suppl 11:139-47. doi: 10.1111/clr.12631. Epub 2015 Jun 13. PMID 26073346
- [Background] Berglundh T, Armitage G, Araujo MG, Avila-Ortiz G, Blanco J, Camargo PM, Chen S, Cochran D, Derks J, Figuero E, Hammerle CHF, Heitz-Mayfield LJA, Huynh-Ba G, Iacono V, Koo KT, Lambert F, McCauley L, Quirynen M, Renvert S, Salvi GE, Schwarz F, Tarnow D, Tomasi C, Wang HL, Zitzmann N. Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S286-S291. doi: 10.1111/jcpe.12957. PMID 29926491
- [Background] Segalla DB, Villarinho EA, Correia ARM, Vigo A, Shinkai RSA. A within-subject comparison of short implants in the posterior region: retrospective study of up to 10 years. J Adv Prosthodont. 2021 Jun;13(3):172-179. doi: 10.4047/jap.2021.13.3.172. Epub 2021 Jun 25. PMID 34234927
- [Background] Villarinho EA, Triches DF, Alonso FR, Mezzomo LAM, Teixeira ER, Shinkai RSA. Risk factors for single crowns supported by short (6-mm) implants in the posterior region: A prospective clinical and radiographic study. Clin Implant Dent Relat Res. 2017 Aug;19(4):671-680. doi: 10.1111/cid.12494. Epub 2017 May 10. PMID 28493384